CLINICAL TRIAL: NCT04086485
Title: Phase I/II Study of Lu-177-DOTATATE (Lutathera) in Combination With Olaparib in Inoperable Gastroenteropancreatico Neuroendocrine Tumors (GEP-NET)
Brief Title: Lu-177-DOTATATE (Lutathera) in Combination With Olaparib in Inoperable Gastroenteropancreatico Neuroendocrine Tumors (GEP-NET)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 190138; 19-C-0138
Record Dates: First submitted 2019-09-10; First posted 2019-09-11 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12-10

CONDITIONS: Gastroenteropancreatico Tumors; Neuroendocrine Tumors; Neuroendocrine Neoplasms
Keywords: Somatostatin Receptors; Peptide receptor radionuclide therapy; Carcinoids; Radionuclide Therapy; olaparib; PARP Inhibitor
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor | interventions — lutetium Lu 177 dotatate; olaparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Lu-177-DOTATATE + Olaparib escalation (Experimental): Lu-177-DOTATATE and escalating doses of olaparib to determine the maximum-tolerated dose (MTD)
  Interventions: Drug: Lu-177-DOTATATE; Drug: Olaparib; Diagnostic Test: Ga dotatate scanning; Diagnostic Test: FDG-PET scanning; Drug: Amino Acid infusion
- 2/Lu-177-DOTATATE + Olaparib fixed dose (Experimental): Lu-177-DOTATATE and olaparib at the MTD
  Interventions: Drug: Lu-177-DOTATATE; Drug: Olaparib; Diagnostic Test: Ga dotatate scanning; Diagnostic Test: FDG-PET scanning; Drug: Amino Acid infusion

INTERVENTIONS:
Drug: Lu-177-DOTATATE — Lu-177-DOTATATE will be given by IV every 8 (+/-2) weeks for a total of 4 administrations
Drug: Olaparib — Olaparib is given as a pill taken orally and is to be taken twice a day, starting from 2 days before the first administration of Lu-177-DOTATATE until 4 weeks after the last administration
Diagnostic Test: Ga dotatate scanning — Ga68-DOTATATE PET/CT scan will be done at baseline, at week 32, then every 24 weeks in followup period.
Diagnostic Test: FDG-PET scanning — F18-FDG PET/CT scan will be done at baseline, at week 32, then every 24 weeks in followup period.
Drug: Amino Acid infusion — Concomitant administration of an IV infusion of an amino acid (AA) solution will also be done for renal protection. The AA infusion will begin at least 30-60 minutes prior to injection of Lu-177-DOTATATE and will continue during and after the Lutathera infusion until the entire prescribed amount is infused.

SUMMARY:
Background:

A neuroendocrine tumor is a rare type of tumor. It comes from body cells called neuroendocrine cells. Sometimes, these tumors develop in the gastrointestinal tract and pancreas. Researchers want to find out if a combination of drugs can shrink these tumors.

Objective:

To learn if people with certain neuroendocrine tumors can take a combination of 2 drugs, Lutathera and Olaparib, without having severe side effects, and if this treatment makes the tumors shrink.

Eligibility:

Adults 18 and older who have a neuroendocrine tumor in the pancreas or intestine that cannot be cured by surgery and has somatostatin receptors on the cells.

Design:

Eligible participants will get Lutathera through an intravenous (IV) infusion every 8 weeks for 4 cycles. One cycle is 8 weeks. Each cycle includes a follow-up visit at week 4. For the IV, a small plastic tube is put into an arm vein.

Participants will also take Olaparib by mouth twice a day for 4 weeks of each cycle. They will use a medicine diary to track the doses.

During the study, participants will have physical exams. They will have blood and urine tests. They will fill out questionnaires about their general well-being and function. Their heart function will be tested. They will have scans of their chest, abdomen, and pelvis. One type of scan will use an IV infusion of a radioactive tracer.

Participants will have a follow-up visit about 4 weeks after treatment ends. Then they will have follow-up visits every 12 weeks for 3 years. Then they will have yearly phone calls.

DETAILED DESCRIPTION:
Background:

* Neuroendocrine tumors (NETs) of the gastrointestinal tract and pancreas are a rare and heterogeneous, but clinically important, group of neoplasms with unique tumor biology, natural history, and clinical management issues.
* While the treatment of localized NETs is surgical resection, a variety of therapeutic options are available for patients with advanced NETs. These include medical control of excess hormone levels and associated symptoms, cytoreductive surgery for patients with advanced disease, radioembolization, chemoembolization, systemic chemotherapy, interferon, longacting somatostatin analogs, receptor-targeted radionuclide therapy, and or liver transplantation.
* Somatostatin receptors (SSTR) have been shown to be overexpressed in a number of human tumors, including neuroblastoma, prostate cancer, pheochromocytomas, paragangliomas, and NETs, among many others.
* Lu-177-DOTATATE (Lutathera) is a SSTR-agonist agent which emits ionizing radiation that causes DNA damage to its target cells through both direct and indirect mechanisms. In addition, ionizing radiation has also been shown to induce cell death through what is known as the bystander effect, a phenomenon where cellular signaling from irradiated cells towards non-irradiated cells induces cellular damage and eventually death in nearby surrounding cells.
* Olaparib is a PARP inhibitor indicated as monotherapy in patients with deleterious or suspected deleterious germline BRCA-mutated advanced ovarian cancer who have been treated with three or more prior lines of chemotherapy. Olaparib has an established safety

profile and it is under investigation in several different cancers.

- The rationale behind using combination therapies in cancer stems from the potential of synergistic mechanisms of action of the involved agents. Olaparib is a PARP-inhibitor which blocks the repair of single-stranded DNA breaks and is especially effective when combined with other agents which induces DNA damage.

Objectives:

* Phase I:

  * Characterize the safety profile and tolerability of the olaparib + Lu-177-DOTATATE combination.
  * Determine the maximum tolerated dose (MTD) dose of the combination using the 3+3 dose escalation design.
* Phase II:

  * Measure the Best Overall Response Rate (BOR) by RECIST 1.1 at the MTD dose at completion of 4 cycles of treatment.

Eligibility:

* Clinical diagnosis of GEP-NET disease, histologically confirmed to be consistent with neuroendocrine tumor.
* Inoperable disease (metastatic, non-candidate for surgery with curative intent, locally advanced into vessels or other critical structures, etc.).
* Age >=18 years.
* Must have presence of SSTR+ disease as documented by positive Ga-68-DOTATATE PET scan within 12 weeks prior to anticipated treatment.
* ECOG Performance Status <= 1.

Design:Design:

* Open-label, single-arm, single-center, phase I/II study evaluating the safety and efficacy of the Lu-177-DOTATATE + olaparib combination in patients with inoperable GEP-NET.
* Each cycle consists of 30 days of olaparib, one infusion of Lu-177 followed by 4 weeks off drug. There will be a total of 4 cycles for each patient, in both phase I and II.
* For the Phase I portion, Lu-177-DOTATATE will be given at the fixed, FDA-approved dose regimen of 200 mCi (7.4 GBq) IV every 8 (+/- 2) weeks for a total of 4 administrations, while olaparib will be evaluated as a radiosensitizer and be dose-escalated from a starting total dose of 100 mg PO up to total dose of 600 mg PO. Administration of olaparib will start 2 days prior to each administration of Lu-177-DOTATATE and will continue daily until 4 weeks after each administration of Lu-177-DOTATATE, and will be restarted 2 days prior to next administration of Lu-177-DOTATATE.
* For the Phase II portion, patients will receive Lu-177-DOTATATE at a fixed dose of 200 mCi (7.4 GBq) in combination with olaparib at the MTD dose as determined in Phase I.
* All patients will be contacted by phone within a week after each Lu-177-DOTATATE treatment for a toxicity assessment. They will also be seen in the NIH clinic every 4 (+/- 1) weeks.
* Approximately 30 days (+/- 1 week) after last dose of study drug, patients will be invited for a safety end of treatment (EOT) visit. After the EOT visit, patients will continue to be invited to NIH CC every 12 weeks until 3 years after the end of treatment visit. Thereafter, all participants will be contacted yearly through any NIH approved platform to assess for disease status.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Clinical diagnosis of GEP-NET disease, histologically consistent with neuroendocrine tumor.
* Inoperable disease (metastatic, non-candidate for surgery with curative intent, locally advanced into vessels or other critical structures, etc.)

NOTE: Presence of at least one non-irradiated index lesion (Phase II only).

* Patients on somatostatin analogue therapy (e.g., but not only limited to sandostatin or lanreotide therapy) must have initiated and been on a consistent dose of therapy for at least 3 months prior to study enrollment.
* Patients on short-term octreotide must have dose held for 24 hours without octreotide because this is necessary for study Lu-177-DOTATATE therapy.
* Age >=18 years. Because no dosing or adverse event data are currently available on the use of Lu-177-DOTATATE in combination with olaparib in patients <18 years of age, children are excluded from this study, but may be eligible for future pediatric trials.
* Must have presence of somatostatin receptors (SSTR) positive disease as documented by positive Ga-68-DOTATATE PET scan within 12 weeks prior to enrollment. NOTE: Positivity of Ga-68-DOTATATE PET scan is defined as having at least one RECIST 1.1 measurable lesion that has an SUV higher than or equal to liver and is qualitatively higher and distinguishable from background activity.
* Known BRCA mutation status (Cohort 3 only).
* Progressive disease by RECIST 1.1, as compared to previous anatomic imaging no more than 36 months from the date of study enrollment, with at least 1 measurable lesion by RECIST 1.1.
* ECOG Performance Status of <=1.
* Patients must have normal organ and bone marrow function measured within 28 days prior to enrollment as defined below:

  * Hemoglobin >= 10.0 g/dL with no blood transfusion in the past 28 days
  * Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
  * Platelet count >= 100 x 10^9/L
  * Total bilirubin <= 1.5 x institutional upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) <= 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be <= 5x ULN
  * Patients must have creatinine clearance estimated of >= 51 mL/min using the Modification of Diet in Renal Disease (MDRD) study equation or based on a 24 hour urine test: eGFR = 175 x (SCr)^-1.154 x (age)^-0.203 x 0.742 [if female] x 1.212 [if Black]
* Ability to understand and willingness to sign informed consent.
* Postmenopausal or evidence of non-childbearing status. For individuals of childbearing potential (IOCBP): negative urine or serum pregnancy test within 28 days of study enrollment. Postmenopausal is defined as:

  * Amenorrheic for 1 year (12 months in a row) or more without an alternative medical cause; if the individual received exogenous hormonal treatments, must be amenorrheic for 1 year or more following cessation of the same
  * Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post-menopausal range for individuals under 50
  * Radiation-induced oophorectomy with last menses >1 year ago
  * Chemotherapy-induced menopause with >1 year interval since last menses
  * Surgical sterilization for IOCBP participants (bilateral oophorectomy or hysterectomy) and/or participants with partners that can bear children.
* NOTE: An individual is not of childbearing potential if a prior history of hysterectomy with bilateral oophorectomy or other procedure has rendered the patient surgically sterile, or >1 years since last menstruation. Must have outside endocrinologist/medical oncologist who can follow the patient for standard of care follow-ups after receiving PRRT at the NIH.
* Study drugs can have adverse effects on embryofetal survival and development. It is further not known whether olaparib or its metabolites are found in seminal fluid. For these reasons:

  * Individuals of childbearing potential and their partners, who are sexually active, must agree to the use of 2 highly effective forms of contraception in combination (male condom plus one of the methods listed below) or must totally/truly abstain from any form of sexual intercourse. This should be started from the signing of the informed consent, throughout study treatment and for at least 7 month for individuals of childbearing potential after the last dose of the study drugs.
  * Patients with partners that can bear children must use a male condom during treatment and for 4 months after the last dose of study drugs when having sexual intercourse with a pregnant individual or with an individual of childbearing potential. Partners of patients should also use a highly effective form of contraception (see below) if they are of childbearing potential. Patients should not donate sperm throughout study treatment and for 4 months following the last dose of study drugs.
  * Acceptable birth control methods include:

    * Total sexual abstinence i.e., refrain from any form of sexual intercourse in line with the patients' usual and/or preferred lifestyle. Abstinence must be for the total duration of the study treatment and for at least 7 months (for IOCBP) or 4 months (for patients with partners of child bearing potential) after the last dose of study treatment. Periodic abstinence (e.g., calendar ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Vasectomised sexual partner PLUS male condom (with participant assurance that partner received post-vasectomy confirmation of azoospermia)
    * Tubal occlusion PLUS male condom
    * Intrauterine Device (provided coils are copper-banded) PLUS male condom
    * Mini pill PLUS male condom: Progesterone-based oral contraceptive pill using desogestrel. Cerazette (Merck Sharp & Dohme) is currently the only highly efficacious progesterone- based pill available
    * Combined pill PLUS male condom: Normal and low-dose combined oral pills
    * Injection PLUS male condom: Medroxyprogesterone injection (eg, Depo-Provera [Pfizer])
    * Implants PLUS male condom: Etonorgestrel-releasing implants (eg, Nexplanon [Merck Sharp & Dohme])
    * Patch PLUS male condom: Norelgestromin/ethinyl estradiol transdermal system (eg, Xulane)
    * Intravaginal device (eg, ethinyl estradiol-/etonogestrel-releasing intravaginal devices such as NuvaRing [Merck Sharp & Dohme]) PLUS male condom
    * Levonorgestrel-releasing intrauterine system (eg, Mirena [Bayer]) PLUS male condom.

EXCLUSION CRITERIA:

* Patients who have any GEP-NET lesions that are negative by Ga-68-DOTATATE-PET imaging but positive by FDG-PET imaging, unless they have progressed on at least one other line of prior systemic treatment (such as chemotherapy or tyrosine kinase inhibitor) and the majority of their tumor lesions are Ga-68-DOTATATE-avid.
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with study drugs, breastfeeding should be discontinued if the mother is treated with study drugs.
* Other known co-existing malignancies except non-melanoma skin cancer and carcinoma in situ of the uterine cervix, unless definitively treated and proven no evidence of recurrence for 5 years.
* Patients who are receiving any other investigational agents.
* Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 4 weeks prior to study enrollment.
* Patients with persistent toxicities (>= CTCAE grade 2) with the exception of alopecia, caused by previous cancer therapy and toxicities deemed irreversible/stable expected to interfere with study drug administration in the opinion of the Principal Investigator.
* Patient's weight exceeding PET table tolerance (> 400 lbs).
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, hypertension (>180/110), arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with symptomatic, uncontrolled brain metastases. NOTE: Patients with previously treated brain metastases are eligible if asymptomatic and may be on a stable dose of corticosteroids as long as these were started at least 4 weeks prior to treatment.
* Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease by imaging and clinical assessment as assessed by the treating investigator for 28 days before enrollment.
* Concomitant use of known strong or moderate CYP3A inhibitors within 2 weeks before enrollment.
* Concomitant use of known strong or moderate CYP3A inducers within 5 weeks (for enzalutamide or phenobarbital) and 3 weeks for other agents before enrollment.
* Patients that have had major surgery within 4 weeks prior to study enrollment and have not recovered from any effects of any major surgery.
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
* Previous allogeneic hematopoietic stem cell transplant, allogeneic bone marrow transplant or double umbilical cord blood transplant (duCBT).
* Patients with a known hypersensitivity to olaparib or Lutathera or any excipients of these products.
* Resting ECG indicating uncontrolled cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, QTcF prolongation >500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome.
* Patients with myelodysplastic syndrome/acute myeloid leukemia or with features suggestive of MDS/AML.
* Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV). HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with study drugs. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Patients with known active hepatitis (i.e., Hepatitis B or C).
* Any previous treatment with PARP inhibitor, including olaparib and/or any previous treatment with any systemic radionuclide agents.
* Involvement in the planning and/or conduct of the study.
* Previous treatment with Lu-177-DOTATATE.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-10-03 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Maximum Tolerated Dose | End of cycle 1
  Depending on what the speed of dose escalation and the final MTD dose, it is estimated that for 4 dose levels with up to 6 patients at each level, approximately 12 to 24 patients will be required for the phase I portion of the study. Standard 3+3 design will be used.
Phase 2: Overall Response Rate | At disease progression
  Proportion of patients who have a partial or complete response to therapy.

SECONDARY OUTCOMES:
Phase 2: PFS and OS of BRCA participants | Disease progression
  Preliminary evidence of exceptional efficacy of the combination at MTD in a sub-cohort of participants with BRCA mutation. Participants from the BRCA cohort will be analyzed together with other phase 2 participants as well as separately using descriptive data only.
Phase 1: BOR and PFS | Disease progression
  Preliminary information on the BOR will be presented as a percentage with 95% confidence intervals. Only evaluate patients will be included. Kaplan-Meier curves of PFS will be constructed. Median PFS will be reported with 95% confidence intervals.
Phase 2: PFS and OS | Death
  Kaplan-Meier curves of PFS and OS will be constructed. Median PFS and OS will be reported with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Frank I Lin, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI. @@@@@@@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Derived] Haque F, Carrasquillo JA, Turkbey EB, Mena E, Lindenberg L, Eclarinal PC, Nilubol N, Choyke PL, Floudas CS, Lin FI, Turkbey B, Harmon SA. An automated pheochromocytoma and paraganglioma lesion segmentation AI-model at whole-body 68Ga- DOTATATE PET/CT. EJNMMI Res. 2024 Nov 5;14(1):103. doi: 10.1186/s13550-024-01168-5. PMID 39500789
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-C-0138.html